CLINICAL TRIAL: NCT03358901
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability and Pharmacokinetics of Multiple Intravenous Administration of YC-6 in Healthy Chinese Adult Subjects
Brief Title: Safety and Pharmacokinetics of Multiple Dose of YC-6 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Cellprotek Pharmaceutical Co., Ltd. (Industry)
Collaborators: Xiuhe Medical Technique Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YC-6-PI-M
Record Dates: First submitted 2016-12-16; First posted 2017-12-02 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- YC-6 (Experimental): 6 volunteers in each level will be infused 100, 200, 400, or 600 mg of YC-6 over 7 consecutive days: BID within 30 minutes for the first 6 days and QD on the 7th day.
  Interventions: Drug: YC-6
- Vehicle (Placebo Comparator): 2 volunteers in each level will be infused 2, 4, 8, or 12 g of vehicle over 7 consecutive days: BID within 30 minutes for the first 6 days and QD on the 7th day.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: YC-6
  Arms: YC-6
Drug: Vehicle
  Arms: Vehicle

SUMMARY:
The study is designed to determine the safety, tolerability, and pharmacokinetics in healthy subjects with multiple intravenous administration of the neuroprotectant YC-6 compared to placebo.

DETAILED DESCRIPTION:
tPA administration within 3-4.5 hours after stroke onset has been the only approved therapy and thus no more than 7% of acute ischemic stroke (AIS) victims worldwide benefited from tPA. A neuroprotectant, YC-6, showed therapeutic effects in preclinical animal models of AIS, indicating its potential as alternative or combined treatment against human AIS.

This randomized, double-blind, placebo-controlled clinical trial is to explore safety and tolerability in healthy Chinese adult volunteers with dose-escalating intravenous infusion of YC-6 for 7 consecutive days. 6 subjects for YC-6 and 2 for placebo will be allocated in each level. Blood and urine samples of each subject will be used in determination of pharmacokinetic properties of the investigational drug.

ELIGIBILITY:
Inclusion Criteria:

1. 18~55 years old healthy subjects
2. BW ≥ 50 kg, BMI 18~28 kg/m²
3. Signed the informed consent from to participate voluntarily and to comply with the trial requirements

Exclusion Criteria:

1. History of clinically significant cardiovascular, hepatic, renal, gastrointestinal, hematologic diseases
2. Clinically significant abnormality evidenced from detailed physical examination, 12-lead ECG, biochemistry, hematology, and routine urine analysis
3. Glomerular filtration rate (GFR) < 80 mL/min
4. Any medication within 2 weeks before the first administration in this study
5. History of clinically significant allergy and hypersensitivity
6. Hepatitis B or C, syphilis, or HIV infection on serological examination
7. History of alcoholic addiction or drug abuse within a year before this study
8. Failing of smoking and drunk cessation (Breath carbon monoxide test > 7 ppm) during this study
9. Participated in any drug trial within 3 months before this study
10. Donated blood or blood product ≥ 400 mL or 2 units within 3 months before this study
11. Dissented to avoid intake of tobacco, alcohol, or caffeine, and strenuous exercise or any behavior that would affect the ADME of YC-6
12. Pregnant or breast-feeding women
13. Other subject conditions unsuitable for enrollment in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience treatment-related adverse events (AEs) and serious adverse events (SAEs) | Day 0 to Day 11
  Any untoward medical events during this study were categorized as severe, moderate, or mild, and related or not related to study treatment.

SECONDARY OUTCOMES:
Plasma Concentration of YC-6 | Day 0 to Day 8
  Concentration of YC-6 in plasma of every subject will be measured during day 0 to day 8.

CONTACTS AND LOCATIONS:
Overall Officials: Bei Hu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No